CLINICAL TRIAL: NCT04811690
Title: Testing the Impact of Front-of-package Claims, Imagery, Nutrition Disclosures, and Added Sugar Warning Labels on Fruit Drinks in an Online Store: A Randomized Controlled Trial
Brief Title: Front-of-package Marketing on Fruit Drinks: Online RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Eric B. Rimm, Professor of Nutrition and Epidemiology, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 76336
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Consumer Behavior; Consumer Preference
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- claim and imagery (Experimental): control condition (status quo) showing a front-of-package (FOP) vitamin C claim and fruit imagery on all fruit-flavored drinks.
  Interventions: Behavioral: front-of-package modification
- imagery only (Experimental): FOP fruit imagery on all fruit-flavored drinks, no vitamin C claim on drinks high in added sugars (>=20 %DV)
  Interventions: Behavioral: front-of-package modification
- claim only (Experimental): FOP vitamin C claim on all fruit-flavored drinks, no fruit imagery on drinks high in added sugars
  Interventions: Behavioral: front-of-package modification
- no claim or imagery (Experimental): No FOP vitamin C claim or fruit imagery on drinks high in added sugars
  Interventions: Behavioral: front-of-package modification
- claim, imagery, and % juice disclosure (Experimental): FOP fruit imagery, vitamin C claim, and % juice disclosure on all fruit-flavored drinks
  Interventions: Behavioral: front-of-package modification
- claim, imagery, and added sugar warning (Experimental): FOP fruit imagery and vitamin C claim on all fruit-flavored drinks; added sugar warning on drinks high in added sugar
  Interventions: Behavioral: front-of-package modification
- claim, imagery, and added sugar warning with teaspoons of added sugar disclosure (Experimental): FOP fruit imagery and vitamin C claim on all fruit-flavored drinks; added sugar warning with teaspoons of added sugar disclosure on drinks high in added sugar
  Interventions: Behavioral: front-of-package modification

INTERVENTIONS:
Behavioral: front-of-package modification — testing front-of-package changes to claims, imagery, disclosures, and added sugar warning labels on fruit-flavored drinks

SUMMARY:
This study will test the independent and combined effects of front-of-package claims, imagery, nutrition disclosures, and added sugar warning labels on parents' purchases and perceptions of beverages for their children.

DETAILED DESCRIPTION:
Fruit drinks are widely consumed by 0-5-year-olds. Parents purchase these drinks for their children in part due to misperceptions that they are healthful, which may be driven by front-of-package (FOP) marketing. The FDA is considering changes to FOP marketing regulations but lacks data on how label elements influence consumer behavior. Our study will test the independent and combined effects of FOP claims, imagery, nutrition disclosures, and added sugar warning labels on parents' purchases and perceptions of beverages for their children.

We will conduct an online randomized controlled trial with 5,000 racially/ethnically diverse primary caregivers of children aged 0-5 years. Participants will choose a beverage for their child in an online store and rate health perceptions of different fruit drinks. Participants will be randomized to see high-added-sugar beverages (>20% DV added sugar/serving) with 1 of 7 FOP label conditions: 1) vitamin C claim and fruit imagery (control); 2) imagery only; 3) claim only; 4) no claim or imagery; 5) claim, imagery, and % juice disclosure; 6) claim, imagery, and added sugar warning; or 7) claim, imagery, and added sugar warning w/teaspoons of added sugar.

Primary outcomes will include total calories and added sugar (grams) from chosen online store beverages. Secondary outcomes will include health perceptions and knowledge of added sugar and % juice content in low- and high-added-sugar fruit drinks.

This research will inform federal regulation to correct health misperceptions of sugary drinks.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child 0-5 years old
* >= 18 years old
* U.S. citizen

Exclusion Criteria:

* Participants who complete the survey in less than 1/3 of the median completion time
* Observations from duplicate IP addresses (keep first observation that is unique)
* Participants who answer data integrity check incorrectly

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5028 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Calories in beverage chosen in online store task | through study completion, an average of 15 minutes
  Calories in beverage chosen in online store task
Added sugar content (grams) of beverage chosen in online store task | through study completion, an average of 15 minutes
  Added sugar content (grams) of beverage chosen in online store task

SECONDARY OUTCOMES:
Percentage of participants that chose a drink high in added sugars in online store task | through study completion, an average of 15 minutes
  Percentage of participants that chose a drink high in added sugars (>=20%DV) in online store task
Percentage of participants that chose each drink category in online store task | through study completion, an average of 15 minutes
  Percentage of participants that chose each drink category (e.g., 100% juice, fruit drinks) in online store task
Fruit drink perceptions: likelihood to purchase for child, how healthy for child, how appealing to child, disease risk perceptions for child | through study completion, an average of 15 minutes
  Fruit drink perceptions: likelihood to purchase for child, how healthy for child, how appealing to child, disease risk perceptions for child
Knowledge of juice and added sugar content in beverage | through study completion, an average of 15 minutes
  Knowledge of % juice and added sugar content (categorical and continuous in grams) in beverage

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rimm, ScD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Online Recruitment, run via Harvard T.H. Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Musicus AA, Roberto CA, Moran AJ, Sorscher S, Greenthal E, Rimm EB. Effect of Front-of-Package Information, Fruit Imagery, and High-Added Sugar Warning Labels on Parent Beverage Choices for Children: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2236384. doi: 10.1001/jamanetworkopen.2022.36384. PMID 36227595